CLINICAL TRIAL: NCT05392595
Title: Effects of Vestibular Rehabilitation Program on Dizziness, Vertigo and Balance in Population With Benign Paroxysmal Vertigo
Brief Title: Effects of Vestibular Rehabilitation Program on Dizziness, Vertigo and Balance in Population With Vertigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/22/0212
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Vertigo
Keywords: Rehabilitation exercises; Vertigo; Balance
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Caw-throne and Cooksey exercise, Epley's repositioning maneuver will be performed also cervical stretches with basic balance exercises.
  Interventions: Other: Cawthrone and cooksey exercises,Epley's repositioning maneuver will be performed also cervical stretches with basic balance exercises.
- Group B (Other): Epley's repositioning maneuver will be performed also cervical stretches with basic balance exercises.
  Interventions: Other: Epley's repositioning maneuver will be performed also cervical stretches with basic balance exercises.

INTERVENTIONS:
Other: Cawthrone and cooksey exercises,Epley's repositioning maneuver will be performed also cervical stretches with basic balance exercises. — Epley "repositioning maneuver will be performed, also cervical stretches and Basic Balance exercises Following Exercises will be performed by patient in next session. Caw-Thorne and Cooksey exercise program. Participants will receive CRM for 6 weeks as needed in each evaluation. Frequency: These exercises will be performed thrice a week on alternate days for 40 min sessions. Post-Intervention Assessment: The patients will be assessed 6 weeks after the beginning of the intervention
  Arms: Group A
Other: Epley's repositioning maneuver will be performed also cervical stretches with basic balance exercises. — Conventional treatment: Epley's repositioning maneuver will be performed also cervical stretches with basic balance exercises.
  Frequency: Participants will receive CRM for 6 weeks as needed in each evaluation. Frequency: These exercises will be performed thrice a week on alternate days for 40 min sessions. Post-Intervention Assessment: The patients will be assessed 6 weeks after the beginning of the intervention
  Arms: Group B

SUMMARY:
Benign Paroxysmal Positional Vertigo (BPPV) is characterized by short, recurrent and intense episodes of vertigo. Repositioning maneuvers have been used for its treatment however, evidence indicated recurrence with these maneuvers. However, the effectiveness of this intervention for improving dynamic and static balance in patients with BPPV is unknown. Vestibular rehabilitation through Caw-throne and Cooksey exercises improves dizziness, balance and gives postural stability. This study aims to determine effects of these exercises in improving the residual symptoms of dizziness and balance impairments after CRM. This randomized controlled trial will recruit patients through convenience sampling. Diagnosed patients of BPPV will be confirmed for inclusion through Dix-Hallpike test. Patients presenting with other neurological, orthopedic or metabolic conditions, patients who have had exposure to any balance exercises or other forms of training that can influence results will also be excluded to limit confounding factors A sample of 26 patients will be taken and divided into two groups each with 13 patients. Group A will receive conventional physical therapy while group B will receive Vestibular Rehabilitation exercises with the conventional physical therapy protocol. The conventional physical therapy protocol will include Cervical stretches and Basic Balance Exercises. The session will be around 40 min on each patient with three session per week on alternate days.The study will evaluate patients through Vertigo symptom Scale (to identify vertigo), Dizziness Handicap Inventory (to identify dizziness),Berg Balance Scale (to identify balance and risk of fall). The data will be analyzed using SPPS software.

DETAILED DESCRIPTION:
Vertigo is the perception of motion, which may be described as a sensation of swaying, tilting, spinning of environment or feeling unbalanced. Due to highly variable descriptions of vertigo, it is often consolidated into the umbrella descriptor 'dizziness', a very common complaint.Vertigo can be of vestibular or peripheral origin or be due to non-vestibular or central causes. Benign paroxysmal positional vertigo (BPPV) is the most common cause of peripheral vertigo, accounting for over half of all cases. One of the treatment options for vestibular disorders (unilateral and bilateral vestibular hypofunction and central or mixed vestibular disorders) is vestibular rehabilitation (VR). This consists of an individualized exercise program which has been developed to address the deficits identified during the physical therapy evaluation and which has been shown to be an effective treatment for patients with dizziness and balance disorders. Currently, this program includes compensatory responses, adaptation for visual-vestibular interaction, substitution and postural control exercises, fall prevention, (re)conditioning activities, and functional retraining.These exercises have been used alone or in conjunction with other vestibular approaches and have been proved effective in improving balance and decreasing fall risk (stroke), postural stability (healthy adults), balance (multiple sclerosis) and decreasing perception of disability (unilateral vestibular hypofunction). Their effectiveness on vertigo, dizziness and balance in patients with BPPV has limited evidence. The current study is designed to determine the effects of Vestibular Rehabilitation exercises on vertigo, dizziness and balance in patients with BPPV. The purpose of this study is that, it will provide the evidence which might improve the treatment strategies for the management of symptoms of BPPV and their recurrence after Canalith Repositioning Maneuver and improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female, Age 30-65 years.

  * BPPV diagnosis confirmed by the: 1. A specific history of vertigo/dizziness evoked by acceleration/deceleration. 2. Symptoms of vertigo during Dix Hallpike Test for Posterior Semicircular canal with or without accompanying nystagmus (objective or subjective BPPV)
  * Patients diagnosed with BPPV for at least 6 months

Exclusion Criteria:

* Central nervous system (CNS) involvement,

  * Meniere's disease,
  * Severe eye disorder, labyrinthitis, vestibular neuritis,
  * Any unstable medical condition (e.g severe hypertension or unstable cardiac diagnosis).
  * Any Cervical pathology.
  * Orthopedic or neurologic diagnoses including sensory loss (e.g diabetes) that might affect postural control and have an impact on functional mobility.

Long-term use of benzodiazepines (more than 20 years).

* Cognitive decline or reduced cultural level that prevents the patient from understanding the assessment, vestibular rehabilitation exercises, and granting informed consent.
* Other Balance Disorders

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Vertigo symptom Scale | 3rd day
  Intensity of visual vertigo in nine challenging situations of visual motions that typically provoke dizziness Internal consistency (Cronbach's alpha: 0.94)
Dizziness Handicap Inventory | 3rd day
  Self-perceived handicapping effects imposed by dizziness. Internal consistency (Cronbach's alpha: 0.92), Test-retest reliability r = 0.95
Berg Balance Scale | 3rd day
  Objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. ICC for total score = 0.988, Testretest reliability r = 0.98

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Ikram, Principal Investigator — Riphah International University
Locations (1):
- Physiotherapy outpatient clinic of Bashir Neuro Institute., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim HJ, Lee JO, Choi JY, Kim JS. Etiologic distribution of dizziness and vertigo in a referral-based dizziness clinic in South Korea. J Neurol. 2020 Aug;267(8):2252-2259. doi: 10.1007/s00415-020-09831-2. Epub 2020 Apr 16. PMID 32300888
- [Background] Pan Q, Zhang Y, Long T, He W, Zhang S, Fan Y, Zhou J. Diagnosis of Vertigo and Dizziness Syndromes in a Neurological Outpatient Clinic. Eur Neurol. 2018;79(5-6):287-294. doi: 10.1159/000489639. Epub 2018 May 24. PMID 29794430
- [Background] You P, Instrum R, Parnes L. Benign paroxysmal positional vertigo. Laryngoscope Investig Otolaryngol. 2018 Dec 14;4(1):116-123. doi: 10.1002/lio2.230. eCollection 2019 Feb. PMID 30828628
- [Background] Yang TH, Xirasagar S, Cheng YF, Wang CH, Lin HC. Increased Risk of Injury Following a Diagnosis of Vertigo: A Population-based Study. Laryngoscope. 2021 Jul;131(7):1633-1638. doi: 10.1002/lary.29519. Epub 2021 Mar 18. PMID 33734445
- [Background] Parker IG, Hartel G, Paratz J, Choy NL, Rahmann A. A Systematic Review of the Reported Proportions of Diagnoses for Dizziness and Vertigo. Otol Neurotol. 2019 Jan;40(1):6-15. doi: 10.1097/MAO.0000000000002044. PMID 30439765
- [Background] Alyono JC. Vertigo and Dizziness: Understanding and Managing Fall Risk. Otolaryngol Clin North Am. 2018 Aug;51(4):725-740. doi: 10.1016/j.otc.2018.03.003. Epub 2018 May 24. PMID 29803531
- [Background] Tramontano M, Consorti G, Morone G, Lunghi C. Vertigo and Balance Disorders - The Role of Osteopathic Manipulative Treatment: A Systematic Review. Complement Med Res. 2021;28(4):368-377. doi: 10.1159/000512673. Epub 2020 Dec 23. PMID 33361695
- [Background] Bressi F, Vella P, Casale M, Moffa A, Sabatino L, Lopez MA, Carinci F, Papalia R, Salvinelli F, Sterzi S. Vestibular rehabilitation in benign paroxysmal positional vertigo: Reality or fiction? Int J Immunopathol Pharmacol. 2017 Jun;30(2):113-122. doi: 10.1177/0394632017709917. Epub 2017 May 9. PMID 28485653
- [Background] Argaet EC, Bradshaw AP, Welgampola MS. Benign positional vertigo, its diagnosis, treatment and mimics. Clin Neurophysiol Pract. 2019 Apr 6;4:97-111. doi: 10.1016/j.cnp.2019.03.001. eCollection 2019. PMID 31193795
- [Background] Concha-Cisternas Y, Guzmán-Muñoz E. Vestibular rehabilitation therapy in elderly with benign paroxysmal positional vertigo. MOJ Gerontol Ger. 2020;5(1):5-8.